CLINICAL TRIAL: NCT03489707
Title: Annual Anal Sampling Using DNA Screening to Identify Men Who Have Sex With Men at Increased Risk for Anal Cancer
Brief Title: The Prevent Anal Cancer Self-Swab Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Cancer Institute (NCI) (NIH); The University of Texas Health Science Center, Houston (Other); M.D. Anderson Cancer Center (Other)
Responsible Party: Principal Investigator, Alan Nyitray, PhD, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: HSC-MS-17-0635; R01CA215403 (NIH)
Record Dates: First submitted 2018-03-29; First posted 2018-04-05 (Actual); Results first posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Anal Cancer
Keywords: anal cancer; human papillomavirus
MeSH Terms: conditions — Anus Neoplasms | interventions — Papillomavirus Vaccines

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based human papillomavirus (HPV) DNA screening (Experimental): Persons randomized to arm 1 will receive an HPV DNA home-based collection kit in the mail at 0 and 12 months.
  Interventions: Behavioral: Home-based human papillomavirus (HPV) DNA screening
- Clinic-based human papillomavirus (HPV) DNA screening (Active Comparator): Persons randomized to arm 2 will attend a clinic where a clinician will collect the DNA specimen at 0 and 12 months.
  Interventions: Behavioral: Clinic-based human papillomavirus (HPV) DNA screening

INTERVENTIONS:
Behavioral: Home-based human papillomavirus (HPV) DNA screening — Persons randomized to arm 1 will receive an HPV DNA home-based collection kit in the mail at 0 and 12 months.
  Arms: Home-based human papillomavirus (HPV) DNA screening
Behavioral: Clinic-based human papillomavirus (HPV) DNA screening — Persons randomized to arm 2 will attend a clinic where a clinician will collect the DNA specimen at 0 and 12 months.
  Arms: Clinic-based human papillomavirus (HPV) DNA screening

SUMMARY:
The purpose of this research study is to find ways to screen for anal cancer among gay, bisexual, and other men who have sex with men (MSM) and transgender persons. This study will try to find out if persons will do annual anal cancer screening, what factors are associated with repeated screening, and how this affects a person's decision to have high-resolution anoscopy.

DETAILED DESCRIPTION:
This is a prospective, randomized, two-arm clinical study to evaluate compliance with annual home-based vs clinic-based DNA screening of anal canal exfoliated cells among Milwaukee HIV+ and HIV- men who have sex with men (MSM) and transgender persons aged ≥25 years. At study entry, persons randomized to arm 1 will receive a home-based collection kit in the mail at 0 and 12 months and those in arm 2 will attend a clinic where a clinician will collect the exfoliated cell specimen at 0 and 12 months. Then, persons will receive high-resolution anoscopy (HRA)-directed biopsy to assess precancerous lesions by study arm. We hypothesize that a majority of persons will comply with annual screening with increased compliance among persons in the home-based arm vs clinic-based arm. The proposed research could indicate that annual HPV DNA screening and subsequent HRA are acceptable to MSM and transgender persons; thus, we will determine how high-risk persons are identified for HRA in light of limited HRA resources. The duration of each participant's activities is expected to be 12 months. The study is expected have participant activity from 2019 to 2023.

ELIGIBILITY:
Inclusion Criteria:

* Be > 25 years of age
* Sex at birth is male or gender identity is a transgender person
* Acknowledge sex with men in the last 5 years, or identify as gay or bisexual
* Understand and be willing to give informed consent
* Be willing to be randomized and able to comply with the protocol
* Spanish and/or English speakers/readers, and
* HIV+ or HIV-

Exclusion Criteria:

* Not acknowledge sex with men in the past five years and not identify as gay or bisexual
* Use of anticoagulants other than Aspirin or NSAIDS
* Prior diagnosis of anal cancer
* Plans to move within 12 months
* Not Milwaukee metro residents
* Not willing to attend one of the designated study clinics at baseline, or
* Inability to give informed consent

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — cis males and transgender persons who have sex with men
Enrollment: 253 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan G Nyitray, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Fully de-identified datasets will be shared with properly trained investigators after assessment of institutional policies, Medical College of Wisconsin Human Protections Committee rules, as well as local, state, and Federal laws and regulations.
Time Frame: Data will become available three years after study completion and be available for five years.
Access Criteria: Fully de-identified datasets will be shared with properly trained investigators after assessment of institutional policies, Medical College of Wisconsin Human Protections Committee rules, as well as local, state, and Federal laws and regulations.

REFERENCES:
- [Derived] Nitkowski J, Giuliano AR, Ridolfi T, Chiao E, Fernandez ME, Schick V, Swartz MD, Smith JS, Nyitray AG. Acceptability of Anal Human Papillomavirus Home Self-Sampling and Clinician Sampling Among Sexual and Gender Minority Individuals in Milwaukee, Wisconsin: The Prevent Anal Cancer Self-Swab Study. LGBT Health. 2024 Jan;11(1):47-56. doi: 10.1089/lgbt.2023.0012. Epub 2023 Oct 24. PMID 37870947
- [Derived] Nyitray AG, Schick V, Swartz MD, Giuliano AR, Fernandez ME, Deshmukh AA, Ridolfi TJ, Ajala C, Brzezinski B, Sandoval M, Nedjai B, Smith JS, Chiao EY. Rationale and design of the Prevent Anal Cancer Self-Swab Study: a protocol for a randomised clinical trial of home-based self-collection of cells for anal cancer screening. BMJ Open. 2021 Jun 29;11(6):e051118. doi: 10.1136/bmjopen-2021-051118. PMID 34187833

RESULTS

PARTICIPANT FLOW:
Period: Baseline
Arm/Group | Home-based Human Papillomavirus (HPV) DNA Screening | Clinic-based Human Papillomavirus (HPV) DNA Screening
Started | 120 | 120
Completed | 107 | 89
Not Completed | 13 | 31
Not completed — These individuals simply did not comply with baseline screening in this compliance study. | 13 | 31
Period: 12 Months
Arm/Group | Home-based Human Papillomavirus (HPV) DNA Screening | Clinic-based Human Papillomavirus (HPV) DNA Screening
Started | 120 (Everyone randomized was invited to participate in the 12-month activities regardless of their compliance with baseline activities; thus, number who started period should not equal the number who completed previous period.) | 120 (Everyone randomized was invited to participate in the 12-month activities regardless of their compliance with baseline activities; thus, number who started period should not equal the number who completed previous period.)
Completed | 78 | 63
Not Completed | 42 | 57
Not completed — These individuals simply did not comply with 12-month screening in this compliance study. | 42 | 57

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Home-based Human Papillomavirus (HPV) DNA Screening | Clinic-based Human Papillomavirus (HPV) DNA Screening | Total
Number analyzed (Participants) | 120 | 120 | 240
Age, Categorical [Count of Participants; unit: Participants] — The unit of analysis is the individual.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 113 | 110 | 223
    >=65 years | 7 | 10 | 17
Age, Continuous [Median (Standard Deviation); unit: years] | 46.5 (13.0) | 44.9 (13.9) | 45.8 (13.4)
Sex/Gender, Customized [Number; unit: participants]
  Man | 115 | 112 | 227
  Trans Man | 0 | 1 | 1
  Trans Woman | 3 | 3 | 6
  Non-binary | 2 | 3 | 5
  Other | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 16 | 31
  Not Hispanic or Latino | 104 | 104 | 208
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 19 | 45
  White | 84 | 91 | 175
  More than one race | 6 | 8 | 14
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 120 | 120 | 240

OUTCOME MEASURES:

1. Primary Outcome: Compliance With Annual Anal HPV DNA Screening
Description: Compliance is assessed by the number of participants who provide specimens for annual anal HPV DNA screening
Time Frame: Baseline
Population: One-hundred and seven of 120 in the Home-Based arm and 89 of 120 in the Clinic-based arm complied at Baseline by providing specimens for annual anal HPV DNA screening (Primary Outcome Measure 1).
Measure: Count of Participants; unit: Participants
Arm/Group | Home-based Human Papillomavirus (HPV) DNA Screening | Clinic-based Human Papillomavirus (HPV) DNA Screening
Number analyzed (Participants) | 120 | 120
Participants
  Provided specimens | 107 | 89
  Did not provide specimens | 13 | 31

2. Primary Outcome: Compliance With Annual Anal HPV DNA Screening
Description: Compliance is assessed by the number of participants who provide specimens for annual anal HPV DNA screening
Time Frame: 12 months
Population: Seventy-eight of 120 in the Home-Based arm and 63 of 120 in the Clinic-based arm complied at 12-months by providing specimens for annual anal HPV DNA screening (Primary Outcome Measure 2).
Measure: Count of Participants; unit: Participants
Arm/Group | Home-based Human Papillomavirus (HPV) DNA Screening | Clinic-based Human Papillomavirus (HPV) DNA Screening
Number analyzed (Participants) | 120 | 120
Participants
  Provided specimens | 78 | 63
  Did not provide specimens | 42 | 57

3. Secondary Outcome: Compliance With Annual Screening Based on HIV Status
Description: The number of participants complying with annual screening with positive or negative HIV status. Compliance is defined as screening at baseline and one year.
Time Frame: 12 months 12 months
Population: The row totals for each column equal the overall number of participants analyzed (the arm totals/column totals).
Measure: Count of Participants; unit: Participants
Arm/Group | Home-based Human Papillomavirus (HPV) DNA Screening | Clinic-based Human Papillomavirus (HPV) DNA Screening
Number analyzed (Participants) | 120 | 120
Participants
  HIV-positive: number analyzed (Participants) | 38 | 27
  HIV-positive: Provided specimens | 27 | 6
  HIV-positive: Did not provide specimens | 11 | 21
  HIV-negative: number analyzed (Participants) | 82 | 93
  HIV-negative: Provided specimens | 51 | 57
  HIV-negative: Did not provide specimens | 31 | 36

4. Secondary Outcome: Compliance With Annual Screening Based on Race/Ethnicity
Description: The number of participants complying with annual screening based on race/ethnicity. Racial and ethnic categories are defined by the NIH as follows: American Indian or Alaska Native, Asian, Black or African American, Hispanic or Latino, Native Hawaiian or Other Pacific Islander, and White.
  Compliance is defined as screening at baseline and one year.
Time Frame: 12 months
Population: The row totals for each column, equal the overall number of participants analyzed (the arm totals/column totals).
Measure: Count of Participants; unit: Participants
Arm/Group | Home-based Human Papillomavirus (HPV) DNA Screening | Clinic-based Human Papillomavirus (HPV) DNA Screening
Number analyzed (Participants) | 120 | 120
Participants
  White/Non Hispanic: number analyzed (Participants) | 76 | 82
  White/Non Hispanic: Provided specimens | 49 | 50
  White/Non Hispanic: Did not provide specimens | 27 | 32
  Black/Non-Hispanic: number analyzed (Participants) | 26 | 19
  Black/Non-Hispanic: Provided specimens | 19 | 6
  Black/Non-Hispanic: Did not provide specimens | 7 | 13
  Hispanic: number analyzed (Participants) | 15 | 16
  Hispanic: Provided specimens | 9 | 6
  Hispanic: Did not provide specimens | 6 | 10
  Asian (Not Hispanic or Latino): number analyzed (Participants) | 1 | 0
  Asian (Not Hispanic or Latino): Provided specimens | 0 | 0
  Asian (Not Hispanic or Latino): Did not provide specimens | 1 | 0
  American Indian/Alaskan Native (Not Hispanic or Latino): number analyzed (Participants) | 0 | 1
  American Indian/Alaskan Native (Not Hispanic or Latino): Provided specimens | 0 | 0
  American Indian/Alaskan Native (Not Hispanic or Latino): Did not provide specimens | 0 | 1
  I don't know/Not Reported: number analyzed (Participants) | 2 | 0
  I don't know/Not Reported: Provided specimens | 1 | 0
  I don't know/Not Reported: Did not provide specimens | 1 | 0
  Other: number analyzed (Participants) | 0 | 2
  Other: Provided specimens | 0 | 1
  Other: Did not provide specimens | 0 | 1

5. Secondary Outcome: Number of Participants Attending High-resolution Anoscopy Based on Race/Ethnicity
Description: The number of participants attending high-resolution anoscopy based on race/ethnicity. Racial and ethnic categories are defined by the NIH as follows: American Indian or Alaska Native, Asian, Black or African American, Hispanic or Latino, Native Hawaiian or Other Pacific Islander, and White.
Time Frame: 12 months
Population: The row totals for each column equal the overall number of participants analyzed (the arm totals/column totals).
Measure: Count of Participants; unit: Participants
Arm/Group | Home-based Human Papillomavirus (HPV) DNA Screening | Clinic-based Human Papillomavirus (HPV) DNA Screening
Number analyzed (Participants) | 120 | 120
Participants
  White/Non-Hispanic: number analyzed (Participants) | 76 | 82
  White/Non-Hispanic: Attended HRA | 41 | 54
  White/Non-Hispanic: Did not attend HRA | 35 | 28
  Black/Non-Hispanic: number analyzed (Participants) | 26 | 19
  Black/Non-Hispanic: Attended HRA | 11 | 8
  Black/Non-Hispanic: Did not attend HRA | 15 | 11
  Hispanic: number analyzed (Participants) | 15 | 16
  Hispanic: Attended HRA | 9 | 7
  Hispanic: Did not attend HRA | 6 | 9
  Asian (Not Hispanic or Latino): number analyzed (Participants) | 1 | 0
  Asian (Not Hispanic or Latino): Attended HRA | 0 | 0
  Asian (Not Hispanic or Latino): Did not attend HRA | 1 | 0
  American Indian/Alaskan Native (Not Hispanic or Latino): number analyzed (Participants) | 0 | 1
  American Indian/Alaskan Native (Not Hispanic or Latino): Attended HRA | 0 | 0
  American Indian/Alaskan Native (Not Hispanic or Latino): Did not attend HRA | 0 | 1
  Other (Not Hispanic or Latino): number analyzed (Participants) | 1 | 2
  Other (Not Hispanic or Latino): Attended HRA | 0 | 2
  Other (Not Hispanic or Latino): Did not attend HRA | 1 | 0
  I don't know/Not reported: number analyzed (Participants) | 1 | 0
  I don't know/Not reported: Attended HRA | 1 | 0
  I don't know/Not reported: Did not attend HRA | 0 | 0

6. Secondary Outcome: Number of Participants Attending High-resolution Anoscopy Based on HIV Status
Description: The number of participants attending high-resolution anoscopy based on positive or negative HIV status.
Time Frame: 12 months
Population: The row totals for each column, equal the overall number of participants analyzed (the arm totals/column totals).
Measure: Count of Participants; unit: Participants
Arm/Group | Home-based Human Papillomavirus (HPV) DNA Screening | Clinic-based Human Papillomavirus (HPV) DNA Screening
Number analyzed (Participants) | 120 | 120
Participants
  HIV-positive: number analyzed (Participants) | 38 | 27
  HIV-positive: Attended HRA | 20 | 12
  HIV-positive: Did not attend HRA | 18 | 15
  HIV-negative: number analyzed (Participants) | 82 | 93
  HIV-negative: Attended HRA | 42 | 59
  HIV-negative: Did not attend HRA | 40 | 34

7. Secondary Outcome: Attendance at High-resolution Anoscopy
Description: Number of participants who attend high-resolution anoscopy (HRA)
Time Frame: 12 months
Population: Sixty-two of 120 home-based participants and 71 of 120 clinic-based participants attended HRA.
Measure: Count of Participants; unit: Participants
Arm/Group | Home-based Human Papillomavirus (HPV) DNA Screening | Clinic-based Human Papillomavirus (HPV) DNA Screening
Number analyzed (Participants) | 120 | 120
Participants
  Attended HRA | 62 | 71
  Did not attend HRA | 58 | 49

8. Other Pre Specified Outcome: Human Papillomavirus (HPV) DNA Persistence and Its Association With High-grade Squamous Intraepithelial Lesions (HSIL).
Description: The number of participants that have DNA persistence at 12 months with and without high-grade squamous intraepithelial lesions (HSIL).
Time Frame: 12 months
Population: Only participants who provided a swab at both baseline and 12 months are assessed for high-risk HPV DNA persistence. Only those assessed for high-risk persistence are included the analysis of the number of high-grade squamous intraepithelial lesions.
Measure: Count of Participants; unit: Participants
Arm/Group | Home-based Human Papillomavirus (HPV) DNA Screening | Clinic-based Human Papillomavirus (HPV) DNA Screening
Number analyzed (Participants) | 120 | 120
Participants
  Attended HRA | 62 | 71
  Assessed for persistence: number analyzed (Participants) | 62 | 71
  Assessed for persistence | 60 | 55
  Persistent: number analyzed (Participants) | 60 | 55
  Persistent | 36 | 17
  persistent ≥HSIL: number analyzed (Participants) | 36 | 17
  persistent ≥HSIL | 14 | 9
  persistent <HSIL: number analyzed (Participants) | 36 | 17
  persistent <HSIL | 22 | 8
  Not persistent: number analyzed (Participants) | 60 | 55
  Not persistent | 24 | 38
  not persistent ≥HSIL: number analyzed (Participants) | 24 | 38
  not persistent ≥HSIL | 3 | 4
  not persistent < HSIL: number analyzed (Participants) | 24 | 38
  not persistent < HSIL | 21 | 34
  Did not attend HRA (preventing HSIL assessment) | 58 | 49

9. Other Pre Specified Outcome: Host/Viral Methylation and Its Association With High-grade Squamous Intraepithelial Lesions.
Description: Mean of host/viral methylation score among participants stratified by high-grade squamous intraepithelial lesions. The Score 5 (S5) methylation score is an arithmetic continuous risk score with a minimum value of 0 and no maximum value. Higher methylation scores indicate higher risk for disease. While a theoretical maximum for a methylation score does not exist, one published maximum value for anal cancer is approximately 100. In this publication (Lorincz et al., Methylation of HPV and a tumor suppressor gene reveals anal cancer and precursor lesions, DOI: 10.18632/oncotarget.17984), a cut-off of 7.5 for methylation score identified all anal cancers and HSIL.
Time Frame: 12 months
Population: Participants who have both high-resolution anoscopy histology result & methylation score (n=133 of 240 total participants) are analyzed here, whether or not they were analyzed for high-risk HPV persistence. Participants who do not have both high-resolution anoscopy biopsy histology result & methylation score = 107 of 240 total participants.
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Total Participants: Participants who have both high-resolution anoscopy biopsy histology result & methylation score (n=133 of 240 total study participants).
- Home-based Human Papillomavirus (HPV) DNA Screening Who Have Both Histology & Methylation Score: Participants who have both high-resolution anoscopy biopsy histology result & methylation score who were also randomized to the home-based arm.
- Clinic-based Human Papillomavirus (HPV) DNA Screening Who Have Both Histology & Methylation Score: Participants who have both high-resolution anoscopy biopsy histology result & methylation score who were also randomized to the clinic-based arm.
Arm/Group | Total Participants | Home-based Human Papillomavirus (HPV) DNA Screening Who Have Both Histology & Methylation Score | Clinic-based Human Papillomavirus (HPV) DNA Screening Who Have Both Histology & Methylation Score
Number analyzed (Participants) | 133 | 63 | 70
scores on a scale
  ≥HSIL: number analyzed (Participants) | 35 | 19 | 16
  ≥HSIL | 6.98 (5.89) | 6.99 (6.70) | 6.96 (4.99)
  <HSIL: number analyzed (Participants) | 98 | 44 | 54
  <HSIL | 3.31 (2.92) | 3.58 (2.97) | 3.10 (2.90)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Home-based Human Papillomavirus (HPV) DNA Screening | Clinic-based Human Papillomavirus (HPV) DNA Screening
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/120
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/120
Other Adverse Events (participants affected / at risk) | 0/120 | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT03489707/Prot_SAP_002.pdf
  • Informed Consent Form (2022-01-03): https://cdn.clinicaltrials.gov/large-docs/07/NCT03489707/ICF_001.pdf